CLINICAL TRIAL: NCT00684476
Title: Maintenance Bee-Venom Immunotherapy Administered at 6-Month Intervals Does Not Protect Against re-Stings
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Meir Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 130504
Record Dates: First submitted 2008-05-21; First posted 2008-05-26 (Estimated); Last update posted 2008-05-26 (Estimated); Status verified 2004-03

CONDITIONS: Venom Allergy
MeSH Terms: conditions — Venom Hypersensitivity | interventions — Desensitization, Immunologic

INTERVENTIONS:
Drug: venom immunotherapy

SUMMARY:
Maintenance venom immunotherapy administered at 6-month intervals to bee-venom allergic patients failed to provide protection from systemic reactions after sting challenges. These patients should continue their immunotherapy at 1-3 month intervals.

DETAILED DESCRIPTION:
Background: The intervals at which maintenance venom immunotherapy (MVIT) is administered have been progressively extended over the years.

Objective: To examine whether the administration of bee venom (BV) maintenance dose (MD) at 6-month interval is safe and efficacious.

Methods: The usual 3-month interval at which venom allergic patients were receiving their MVIT was gradually extended to 6 months. Systemic reactions (SRs) to immunotherapy injections or to field stings were regularly recorded. BV allergic patients were deliberately sting-challenged after reaching the 6-month interval.

ELIGIBILITY:
Inclusion Criteria:

* Venom allergy

Exclusion Criteria:

* none

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2004-06; Study Completion 2006-05

PRIMARY OUTCOMES:
whether the administration of bee venom (BV)
maintenance dose (MD) at 6-month interval is safe and
efficacious.

CONTACTS AND LOCATIONS:
Overall Officials: Arnon Goldberg, M.D, Principal Investigator — The Allergy and Clinical Immunology Unit, Meir Hospital, Kfar-Saba, Israel, affiliated with The Sackler School of Medicine, Tel-Aviv University, Tel-Aviv, Israel